CLINICAL TRIAL: NCT04891991
Title: Treatment of Proliferative Vitreoretinopathy With Intravitreal Infliximab
Brief Title: Intravitreal Infliximab for Proliferative Vitreoretinopathy
Acronym: FIXER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Gehad Elnahry, Lecturer of Ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU272021
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Rhegmatogenous Retinal Detachment; Proliferative Vitreoretinopathy; Retinal Detachment
MeSH Terms: conditions — Vitreoretinopathy, Proliferative; Retinal Detachment | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Infliximab group (Active Comparator): This group will receive 1 mg/0.05 mL of intravitreal infliximab at the end of standard pars plana vitrectomy.
  Interventions: Drug: Intravitreal infliximab; Procedure: Pars plana vitrectomy
- Standard of care group (Sham Comparator): This group will undergo standard pars plana vitrectomy.
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Drug: Intravitreal infliximab — 1 mg/0.05 mL of infliximab will be injected intravitreally at the end of pars plana vitrectomy.
  Other Names: Remicade
  Arms: Infliximab group
Procedure: Pars plana vitrectomy — Standard pars plana vitrectomy

SUMMARY:
Proliferative vitreoretinopathy (PVR) is the most common cause for failure of rhegmatogenous retinal detachment repair and is characterized by the growth and contraction of cellular membranes within the vitreous cavity on both sides of the retinal surface as well as intraretinal fibrosis.

Multiple therapeutic agents have been tried as an adjunctive to retinal detachment surgery for PVR with no consistent efficacy. Tumor necrosis factor-α (TNF-α), which is a prominent inflammatory cytokine, is secreted in response to trauma, infection, and inflammation. It is a key mediator of ocular inflammation and its interactions with the retinal pigment epithelium (RPE) cell contribute to the initiation of PVR. This may occur through the action of TNF-α on the RPE cells inducing changes in cellular morphologies that lead to the formation of fibroblastic cells.

Infliximab (Remicade; Janssen Biotech, Horsham, PA, USA) is a mouse-human chimeric antibody that neutralizes the biological activity of TNF-α by high-affinity binding to the soluble and transmembrane forms of TNF-α, therefore preventing the effective binding of TNF-α with its receptors. Infliximab is used in the treatment of various ocular and systemic inflammatory conditions. Furthermore, intravitreal infliximab has been used for the treatment of various ocular diseases and has proven to be generally safe for the short term in inflammatory ocular conditions. A recent study showed that intravitreal infliximab can inhibit the development of PVR and reduce levels of cytokines in an experimental dispase-induced PVR model.

The purpose of this randomized controlled trial is to evaluate the efficacy of intravitreal infliximab injection as an adjunct to pars plana vitrectomy in the treatment of PVR associated with primary rhegmatogenous retinal detachment.

DETAILED DESCRIPTION:
Proliferative vitreoretinopathy (PVR) is the most common cause for failure of rhegmatogenous retinal detachment repair and is characterized by the growth and contraction of cellular membranes within the vitreous cavity on both sides of the retinal surface as well as intraretinal fibrosis.

The incidence of PVR in all cases of retinal detachment is estimated to be 5- 10%. The incidence of PVR has largely remained unchanged in prospective studies despite the evolution of vitreoretinal techniques over the past 25 years, including valved trocars and smaller gauge instrumentation.

Numerous risk factors for the development of PVR have been identified. Almost all risk factors for PVR are associated with intravitreal dispersion of retinal pigment epithelial cells or breakdown of the blood-ocular barrier. Following a retinal break, the retinal pigment epithelial (RPE) cells are exposed to the vitreous cavity to react to growth factors and cytokines in the vitreous, resulting in a forward feedback to secret more growth factors and cytokines to further stimulate cellular responses.

Multiple therapeutic agents have been tried as an adjunctive to retinal detachment surgery for PVR with no consistent efficacy. Tumor necrosis factor-α (TNF-α), which is a prominent inflammatory cytokine, is secreted in response to trauma, infection, and inflammation. It is a key mediator of ocular inflammation and its interactions with RPE cells contribute to the initiation of PVR. This is because TNF-α was found to act on the RPE cells consequently inducing changes in cellular morphologies leading to the formation of fibroblastic cells. Additionally, if TNF-α is combined with other growth factors, a strong synergistic effect can be induced to form epithelial-mesenchymal transition (EMT)-associated fibrotic focus.

Infliximab (Remicade; Janssen Biotech, Horsham, PA, USA) is a mouse-human chimeric antibody that neutralizes the biological activity of TNF-α by high-affinity binding to the soluble and transmembrane forms of TNF-α, therefore preventing the effective binding of TNF-α with its receptors. Infliximab is used in the treatment of various ocular and systemic inflammatory conditions. Furthermore, intravitreal infliximab has been used for the treatment of various ocular diseases and has proven to be generally safe for the short term in inflammatory ocular conditions. A recent study showed that intravitreal infliximab can inhibit the development of PVR and reduce levels of cytokines in an experimental dispase-induced PVR model.

The purpose of this randomized controlled trial is to evaluate the efficacy of intravitreal infliximab injection as an adjunct to pars plana vitrectomy in the treatment of PVR associated with primary rhegmatogenous retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than or equal to 18 years
* Primary rhegmatogenous retinal detachment with proliferative vitreoretinopathy more than or equal to grade C

Exclusion Criteria:

* Patients with a history of open globe injury
* Recurrent retinal detachment or primary failed retinal detachment surgery
* History of vitreoretinal procedure
* Retinal vascular diseases (Diabetic retinopathy, retinal vein occlusion,...etc)
* Pregnant or breastfeeding females
* Inability to attend regular follow-up visits
* History of pulmonary or extra-pulmonary tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Anatomical success | 9 months
  Anatomical Success will be defined as stable complete retinal reattachment following pars plana vitrectomy and silicone oil removal.

SECONDARY OUTCOMES:
Visual acuity | 1, 3, 6, and 9 months
  Best corrected visual acuity will be measured at follow up visits using standard Snellen charts.
Macular structure | 1, 3, 6, and 9 months
  Optical coherence tomography will be done at each follow up visit to assess the structure of the macula.
Macular vascularity | 7 months
  Optical coherence tomography angiography will be done at each follow up visit to assess macular vascular density.
Macular function | 7 months
  Macular function will be assessed during follow up visits using multifocal electroretinography
Single operation success rate | 9 months
  The rate of successful retinal reattachment following a single operation will be calculated.
Recurrence rate | 9 months
  Cumulative rate of recurrence of retinal detachment and reoperation following the primary surgery will be calculated during the study period.
Epiretinal proliferative | 1, 3, 6, and 9 months
  The formation of significant epiretinal proliferation will be assessed clinically at each follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman G Elnahry, MD, PhD, Principal Investigator — Cairo University; Hany S Hamza, MD, PhD, Study Chair — Cairo University; Ahmed M Younes, MD, MSc, Principal Investigator — Cairo University; Ahmed A Abdel-Kader, MD, PhD, Study Director — Cairo University; Ahmed M Abdelbaki, MD, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagasaki H, Shinagawa K, Mochizuki M. Risk factors for proliferative vitreoretinopathy. Prog Retin Eye Res. 1998 Jan;17(1):77-98. doi: 10.1016/s1350-9462(97)00007-4. PMID 9537796
- [Background] Pastor JC. Proliferative vitreoretinopathy: an overview. Surv Ophthalmol. 1998 Jul-Aug;43(1):3-18. doi: 10.1016/s0039-6257(98)00023-x. PMID 9716190
- [Background] Pastor JC, de la Rua ER, Martin F. Proliferative vitreoretinopathy: risk factors and pathobiology. Prog Retin Eye Res. 2002 Jan;21(1):127-44. doi: 10.1016/s1350-9462(01)00023-4. PMID 11906814
- [Background] Pennock S, Haddock LJ, Mukai S, Kazlauskas A. Vascular endothelial growth factor acts primarily via platelet-derived growth factor receptor alpha to promote proliferative vitreoretinopathy. Am J Pathol. 2014 Nov;184(11):3052-68. doi: 10.1016/j.ajpath.2014.07.026. Epub 2014 Sep 26. PMID 25261788
- [Background] Charteris DG, Sethi CS, Lewis GP, Fisher SK. Proliferative vitreoretinopathy-developments in adjunctive treatment and retinal pathology. Eye (Lond). 2002 Jul;16(4):369-74. doi: 10.1038/sj.eye.6700194. PMID 12101443
- [Background] Leiderman YI, Miller JW. Proliferative vitreoretinopathy: pathobiology and therapeutic targets. Semin Ophthalmol. 2009 Mar-Apr;24(2):62-9. doi: 10.1080/08820530902800082. PMID 19373688
- [Background] Heimann H, Bartz-Schmidt KU, Bornfeld N, Weiss C, Hilgers RD, Foerster MH; Scleral Buckling versus Primary Vitrectomy in Rhegmatogenous Retinal Detachment Study Group. Scleral buckling versus primary vitrectomy in rhegmatogenous retinal detachment: a prospective randomized multicenter clinical study. Ophthalmology. 2007 Dec;114(12):2142-54. doi: 10.1016/j.ophtha.2007.09.013. PMID 18054633
- [Background] Savur F, Aydemir O, Ilhan N. The effect of infliximab and octreotide on cytokine levels experimental proliferative vitreoretinopathy. Cutan Ocul Toxicol. 2020 Mar;39(1):61-66. doi: 10.1080/15569527.2019.1701000. Epub 2019 Dec 17. PMID 31809602
- [Background] Markomichelakis N, Delicha E, Masselos S, Sfikakis PP. Intravitreal infliximab for sight-threatening relapsing uveitis in Behcet disease: a pilot study in 15 patients. Am J Ophthalmol. 2012 Sep;154(3):534-541.e1. doi: 10.1016/j.ajo.2012.03.035. Epub 2012 Jul 11. PMID 22789563
- [Background] Pascual-Camps I, Hernandez-Martinez P, Monje-Fernandez L, Dolz-Marco R, Gallego-Pinazo R, Wu L, Arevalo JF, Diaz-Llopis M. Update on intravitreal anti-tumor necrosis factor alpha therapies for ocular disorders. J Ophthalmic Inflamm Infect. 2014 Oct 15;4:26. doi: 10.1186/s12348-014-0026-8. eCollection 2014. PMID 25825604
- [Background] Pastor JC, Rojas J, Pastor-Idoate S, Di Lauro S, Gonzalez-Buendia L, Delgado-Tirado S. Proliferative vitreoretinopathy: A new concept of disease pathogenesis and practical consequences. Prog Retin Eye Res. 2016 Mar;51:125-55. doi: 10.1016/j.preteyeres.2015.07.005. Epub 2015 Jul 21. PMID 26209346
- [Background] Hamza MM, Macky TA, Sidky MK, Ragab G, Soliman MM. INTRAVITREAL INFLIXIMAB IN REFRACTORY UVEITIS IN BEHCET'S DISEASE: A Safety and Efficacy Clinical Study. Retina. 2016 Dec;36(12):2399-2408. doi: 10.1097/IAE.0000000000001109. PMID 27870802
- [Background] Korthagen NM, van Bilsen K, Swagemakers SM, van de Peppel J, Bastiaans J, van der Spek PJ, van Hagen PM, Dik WA. Retinal pigment epithelial cells display specific transcriptional responses upon TNF-alpha stimulation. Br J Ophthalmol. 2015 May;99(5):700-4. doi: 10.1136/bjophthalmol-2014-306309. Epub 2015 Feb 13. PMID 25680620
- [Background] Pennock S, Haddock LJ, Eliott D, Mukai S, Kazlauskas A. Is neutralizing vitreal growth factors a viable strategy to prevent proliferative vitreoretinopathy? Prog Retin Eye Res. 2014 May;40:16-34. doi: 10.1016/j.preteyeres.2013.12.006. Epub 2014 Jan 9. PMID 24412519